CLINICAL TRIAL: NCT06132230
Title: Potential Value of Immunohistochemical Expression of SOX17 and E-Cadherin in Variable Endometrial Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Gehad Bahgat Abdelhameed, Assistant lecturer of Pathology, Sohag University
Other Study IDs: Soh-Med-10-11MD
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Variable Endometrial Lesions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrial carcinoma (EC) is the 6th most commonly occurring cancer in women and the 15th most common cancer overall According to facts derived from Globocan for the year 2020.The overall incidence was 417,367 and 97,370 died due to it. There were more than 417,000 new cases of endometrial cancer in 2020 .EC incidence is predicted to continue to rise in the coming decades, in particular among low and middle-income countries.

SOX17 protein (SRY-box 17) is a member of the SRY-related HMG-box (SOX) family of transcription factors that controls the first step of gene expression and regulates cellular growth and differentiation in the endoderm, during hematopoiesis, and in the cardiovascular system E-Cadherin is a calcium-dependent cell adhesion protein (predicted molecular weight of 97 kDa) that plays a vital role in cell migration and proliferation. The E-cadherin epithelial cell adhesion protein is a tumor suppressor that has an important role in tumor metastasis The loss of expression of E-Cadherin during the epithelial mesenchymal transition (EMT) is often thought to promote metastasis by allowing the dissociation and invasion of cancer cells

The aim of this study is:

1. To evaluate accuracy of SOX17 expression in neoplastic and hyperplastic endometrial lesions.
2. To correlate SOX17 expression with some clinical and pathological parameters of endometrial carcinoma.
3. To evaluate E-Cadhrin expression and its relation to SOX17 in neoplastic and hyperplastic lesions

ELIGIBILITY:
Inclusion Criteria:

* 1. Specimens of total abdominal hysterectomy and bilateral salpingio-oopherectomy of endometrial carcinoma patients 2. D&C of endometrial tissue suspected of hyperplastic or neoplastic lesions

Exclusion Criteria:

* • Specimens with insufficient clinical data.

  * Specimens with extensive necrosis

Ages: 25 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Formalin-fixed paraffin blocks from 70 patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Potential Value of Immunohistochemical Expression of SOX17 and E-Cadherin in Variable Endometrial Lesions | one or two days after staining sections with markers
  Immunohistochemical expression of SOX17 and E-Cadherin in Variable Endometrial Lesions

CONTACTS AND LOCATIONS:
Overall Officials: Gehad Bahgat, Principal Investigator — Sohag faculty of Medicine
Locations (1):
- Sohag faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided